CLINICAL TRIAL: NCT06495346
Title: Identification and Characterisation of Sleep Disorders in a Population of Patients With Non-small Cell Lung Cancer
Acronym: SomOncoP
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9002
Record Dates: First submitted 2024-02-13; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-02

CONDITIONS: Cell Lung Cancer; Sleep Disorders
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: self-questionnaires exploring — At each stage, subjects are asked to fill in self-questionnaires exploring the quality of their sleep, their potential distressing symptoms, their psychological state and the quality of their life at that moment. They complete the self-questionnaires at t

SUMMARY:
This exploratory study will identify and characterise disorders frequently reported by patients as contributing to or altering their quality of life. This will enable a decision tree to be drawn up for diagnosis, referral and treatment of the sleep disorders collected, tailored to patients in this population.

This decision tree should help to improve the management of patients with a cancer diagnosis presenting with sleep disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 and over.
* Being monitored and treated for non-small cell lung cancer.
* With or without ongoing cancer-specific treatment. With no neurocognitive impairment (MoCA test score ≥26/30).
* With a clinically assessed life expectancy of more than 3 months (Royal Marsden Hospital 0-1) and general health (ECOG <2).
* Able to understand the study documents written in French
* Able to complete the study questionnaires written in French.
* Contactable by telephone throughout the study
* Affiliated to a social security scheme or entitled beneficiary
* Not opposed to taking part in the study

Exclusion Criteria:

* Patient refusing to take part in the study
* With a mental illness of the psychosis type monitored and treated prior to the study
* Patient under guardianship or curatorship
* Patient under court protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of non-small cell lung cancer followed and treated by the Oncopneumology Department of the Nouvel Hôpital Civil in Strasbourg
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2025-04-11 (Estimated); Study Completion 2025-06-11 (Estimated)

PRIMARY OUTCOMES:
Score sleep quality criteria (Pittsburgh Sleep Quality Index) | Every 14 days for 2 months
  The overall score ranging from 0 to 21 points. A score of 0 means that there is no difficulty sleeping, and 21 indicates, on the contrary, major difficulties.

CONTACTS AND LOCATIONS:
Locations (1):
- HUS, Strasbourg, Grand Est, France